CLINICAL TRIAL: NCT04471740
Title: Normal-pressure Hydrocephalus. Relationship Between Sleep Apnea and Intracranial and Intraabdominal Pressures. Outcome Prognostic Factors in CSF Shunting. Features Guiding to Implant a Ventricle-peritoneal Versus a Ventriculo-atrial Shunt
Brief Title: Normal Pressure Hydrocephalus and Sleep Apnea
Acronym: NPH/OSA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Valencia (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 2020-07-02
Record Dates: First submitted 2020-07-03; First posted 2020-07-15 (Actual); Last update posted 2022-11-03 (Actual); Status verified 2022-07

CONDITIONS: Normal Pressure Hydrocephalus; Sleep Apnea; Cerebrospinal Fluid Shunt Occlusion
Keywords: Normal pressure hydrocephalus; Sleep apnea; CSF shunt diversion; Ventriculo-peritoneal shunt; Ventriculo-atrial shunt
MeSH Terms: conditions — Hydrocephalus, Normal Pressure; Sleep Apnea Syndromes

STUDY DESIGN:
Intervention Model Description: Patients diagnosed of normal-pressure hydrocephalus will undergo sleep studies to rule our sleep apnea. Those with sleep apnea will be treated for this condition and we will see if the hydrocephalus symptoms improve
Who Masked: Participant
Masking Description: Patients will not be informed of the final treatment decided
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Normal-pressure hydrocephalus only (Experimental): Patients suffering from normal-pressure hydrocephalus with NO sleep apnea
  Interventions: Procedure: CSF shunt diversion
- Normal-pressure hydrocephalus with sleep apnea (Active Comparator): Patients suffering from normal-pressure hydrocephalus with sleep apnea
  Interventions: Procedure: CSF shunt diversion

INTERVENTIONS:
Procedure: CSF shunt diversion — Clinical response to a CSF shunt insertion

SUMMARY:
Normal-pressure hydrocephalus is associated with increases in the intracranial pressure during the night sleep. Sleep apnea also increases the intracranial pressure during the apneic spells. When patients are operated the distal part of the shunt is inserted inside the abdominal cavity, which pressure also increases during the sleep apnea episodes. this is particularly important considering that the recumbent position used to sleep further increases the intraabdominal pressure and that impairs the CSF drainage through the shunt system. The purpose of this study is to analyze the intracranial and intraabdominal pressures during the sleep, particularly during the sleep apnea episodes to see which shunt should be used, to which cavity should be drained (peritoneum or heart) and if correcting the sleep apnea has some positive result on the hydrocephalus symptoms.

DETAILED DESCRIPTION:
Chronic hydrocephalus in adults, also known as normal pressure hydrocephalus or normal pressure hydrocephalus, occurs with the classic Hakim-Adams triad, gait ataxia, or "magnetic gait", urinary incontinence and dementia.

Most of the cases have an idiopathic origin and are the only potentially reversible cause of dementia with surgical treatment (by shunting the cerebrospinal fluid or CSF from the lateral ventricles or the thecal sac to the peritoneal cavity or the right atrium), so it is especially important to diagnose it and treat it properly.

Unfortunately, and despite all the diagnostic arsenal, the results of treatment using cerebrospinal fluid shunts (lumbo-peritoneal or ventricle-peritoneal), even in the best series, show 20-25% of poor results. These poor results have been attributed to many factors, including associated cerebral vascular pathology problems, co-existing dementia symptoms not always well diagnosed, Parkinson's disease, and, lastly, alterations in ventilatory rhythm. during the night, specifically obstructive sleep apnea or OSA.

In reality, the name of normotensive hydrocephalus or hydrocephalus at normal pressure is inaccurate because the intracranial pressure does rise and very markedly during sleep, particularly during the REM phase of sleep. What is no longer so well known is because of such significant increases in intracranial pressure occur. One possible explanation would be that obstructive sleep apnea causes increased intracranial pressure. But it remains to be clarified whether all patients with adult chronic hydrocephalus have sleep apnea, the mechanism of action, and to what extent the treatment of hydrocephalus acts on sleep apnea and vice versa.

Another aspect to consider is that the cerebrospinal fluid shunts work by the pressure gradient between the intracranial cavity and the cavity into which the cephalo-spinal fluid is drained66, usually the peritoneal fluid. During sleep apnea, there should be an increase in intra-abdominal pressure, which would result in the ventricle-peritoneal and lumbo-peritoneal shunts working suboptimally precisely at the time of day when they are most needed, that is when intracranial pressure increases. But this correlation has never been investigated or at least there are no publications about it.

Therefore, it is necessary to know the relationship between intracranial pressure, sleep apnea, and intra-abdominal pressure at night. With these data, it will be possible to better understand the dynamics of the circulation of the cerebrospinal fluid during the night (when it is more pathological in chronic hydrocephalus in adults), what type of bypass valve is the most indicated (whether or not it must have an anti-system siphon if it must be a gravitational or flow valve) and in which patients the implantation of a ventricle-atrial shunt may be an option to consider.

ELIGIBILITY:
Inclusion Criteria:

* Clinical condition compatible with normal-pressure hydrocephalus

Exclusion Criteria:

* Cerebral vascular disease
* Dementia not due to normal-pressure hydrocephalus
* Parkinson's disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-07-02 (Actual); Primary Completion 2023-07-02 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Change of hydrocephalus symptoms with Mini-Mental State Examination | 1-2 months
  Patients will be evaluated with the Mini_mental State Examination before and after CSF shunting to see the degree of improvement they get from this surgical treatment
Change of hydrocephalus symptoms with NPH scale after CSF shunt diversion | 1-2 months
  Patients will be evaluated with the NPH before and after CSF shunting to see the degree of improvement they get from this surgical treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Vicente Vanaclocha, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kawada T. Obstructive sleep apnea in patients with idiopathic normal-pressure hydrocephalus. J Neurol Sci. 2019 Feb 15;397:155. doi: 10.1016/j.jns.2019.01.006. Epub 2019 Jan 10. No abstract available. PMID 30640151